CLINICAL TRIAL: NCT05840822
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study Evaluating the Efficacy and Safety of CBD TPM Capsules in Adults for Use in the Reduction of Insomnia Severity
Brief Title: Evaluating Efficacy and Safety of CBD TPM Capsules for Use in Insomnia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Avecho Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVE047-22
Record Dates: First submitted 2023-04-23; First posted 2023-05-03 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-04

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cannabidiol; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Nightly dose of two placebo capsules
  Interventions: Drug: Placebo
- 75mg CBD (Experimental): Nightly dose of one 75mg CBD capsule and one placebo capsule
  Interventions: Drug: Cannabidiol (CBD) Capsule 75mg; Drug: Placebo
- 150mg CBD (Experimental): Nightly dose of two 75mg CBD capsules
  Interventions: Drug: Cannabidiol (CBD) Capsule 75mg

INTERVENTIONS:
Drug: Cannabidiol (CBD) Capsule 75mg — Cannabidiol (CBD) capsule containing 75mg CBD
  Arms: 150mg CBD; 75mg CBD
Drug: Placebo — Placebo capsule without cannabidiol
  Arms: 75mg CBD; Placebo

SUMMARY:
Insomnia is a common sleep disorder in which a person has difficulty falling asleep or staying asleep or getting good quality sleep. Consequences of insomnia include daytime sleepiness, poor memory function, decline in concentration with negative impacts on social and work activities. Although medical cannabis and cannabis products are widely used worldwide for the management of symptoms associated with insomnia, there is little clinical data available to support the efficacy or utility of CBD in the management of sleep disorders. The proposed study will assess whether nightly doses of 75mg or 150mg of an 8 week period are able to improve patient reported sleep quality when compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 years or older at the time of informed consent.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Provide a signed and dated patient information and consent form (PICF) for the study.
4. Met the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for insomnia disorder, as follows:

   * Complained of dissatisfaction with night-time sleep in the form of difficulty getting to sleep, difficulty staying asleep and/or awakening earlier in the morning than desired despite adequate opportunity for sleep.
   * Frequency of the complaint ≥3 times per week.
   * Duration of complaint ≥3 months.
   * Associated with a complaint of daytime impairment.
5. History of subjective Sleep Onset Latency (sSOL) ≥30 minutes on at least 3 nights per week in the previous 4 weeks AND/OR subjective Wake After Sleep Onset (sWASO) ≥30 minutes on at least 3 nights per week in the previous 4 weeks.
6. Subject reports a regular time spent in bed, either sleeping or trying to sleep is between 7-10 hours.
7. Subjects must have clinical insomnia symptoms as classified by an insomnia severity index (ISI) Score of ≥15.
8. Confirmation of current insomnia symptoms as determined from the Sleep Diary completed on at least 7 consecutive mornings (minimum 5 of 7 for eligibility), such that sSOL ≥30 minutes on at least 3 of the 7 nights and/or sWASO ≥30 minutes on at least 3 of the 7 nights.
9. Subject reports a typical bedtime, (defined as the time the subject attempts to sleep), between 21:00 and 01:00, and waketime, (defined as the time the subject got out of bed for the day), between 05:00 and 10:00.
10. Subject has access to and is able to use a smart phone.
11. Female subjects of childbearing potential must be abstinent or agree to use a highly effective method of contraception for 30 days prior to Day 1, during the study, and for at least 28 days following the last dose of Investigational Product (IP). Agrees to refrain from donating eggs (ova, oocytes) (from Day 1 until 28 days following the last dose of IP).
12. Male subjects that are not surgically sterile (i.e., vasectomy) must be abstinent or agree to use effective barrier contraception (i.e., condom) from Day 1 and for at least 28 days following the last dose of IP and agrees to refrain from sperm donation (from Day 1 until 28 days following the last dose of IP).

Exclusion Criteria:

1. Significant insomnia caused during another sleep-wake disorder, including narcolepsy, a breathing-related sleep disorder, a circadian rhythm sleep-wake disorder, a parasomnia, restless leg syndrome, or an exclusionary score on the Sleep Disorders Screening Battery, or Epworth Sleepiness Scale score as follows:

   * STOP-Bang score ≥5.
   * International Restless Legs Scale score ≥16.
   * Epworth Sleepiness Scale score >15 (scores of 11-15 required excessive daytime sleepiness to be recorded in subject's medical history).
2. Reports symptoms potentially related to narcolepsy that in the clinical opinion of the Investigator indicates the need for referral for a diagnostic evaluation for the presence of narcolepsy.
3. Reports a history of sleep-related violent behavior, or sleep driving, or any other complex sleep-related behavior, e.g., making phone calls, or preparing and eating food while asleep.
4. Beck Depression Inventory - (BDI II) score >19 at Screening.
5. Beck Anxiety Inventory >15 at Screening.
6. Habitually napped more than three times per week.
7. Current or recent cannabis use, within 30 days of consent, and throughout the study.
8. Use of any drug known to affect sleep, within 30 days of Screening and throughout the study, including:

   * Sedatives (e.g. benzodiazepines, zopiclone, eszopiclone, zaleplon, zolpidem, agomelatine, suvorexant, dual orexin receptor antagonists, sodium oxybate mirtazipine (sedating SSRI) and all tricyclic antidepressants,, , sedating H antihistamines (cyproheptadine, dexchlorpheniramine, promethazine, trimeprazine, doxylamine, diphenhydramine, cyclizine),, antipsychotics, melatonin, valerian).
   * Opioids (e.g. morphine, codeine, oxycodone, methadone, buprenorphine, fentanyl, tramadol, tapentadol, hydromorphone).
   * Stimulants (e.g. modafinil, methylphenidate, dexamphetamine, phentermine).
9. Have care responsibilities for an infant <1 year of age.
10. Females who are pregnant or lactating.
11. Have excessive caffeine use (>300 mg or ~3 cups of caffeinated beverages a day) that, in the opinion of the Investigator, contributes to the subject's insomnia, and is unwilling to forgo caffeine-containing beverages for the duration of their participation in the study. Any caffeine consumed needs to be prior to 4:00 pm.
12. PI determined excessive history of acute or severe bronchial asthma (excluding childhood or exercise induced asthma), diagnosed obstructive sleep apnea, hypoxia, hypoxemia, hypercarbia, or other obstructive airway disease or any condition that may increase the risk for respiratory depression.
13. History of neurologic conditions such as seizures or convulsive disorders (including epilepsy), severe head injury or increased intracranial pressure.
14. A calculated creatinine clearance of < 85 mL/minute at Screening according to the equation using Cockcroft and Gault.
15. Liver function tests for alanine transaminase or aspartate aminotransferase > 1.5 times the upper limit of normal at Screening.
16. History of clinically significant (in the opinion of the Investigator) other cardiovascular, pulmonary, neurologic or renal disorders or hepatic, gastrointestinal, oral (difficulty swallowing / taking oral medication), hematological, endocrine, or psychiatric impairment/disorders.
17. Use of any over the counter product, or other medicine derived from hemp or containing cannabidiol, within 30 days of Screening and for duration of study.
18. Known intolerance, allergy or hypersensitivity reactions to cannabis or cannabinoid products (e.g. hemp), and excipients of the IP.
19. Currently taking or have taken drugs that are moderate or strong inhibitors of CYP3A4 or CYP2C19 within 2 weeks or 5 half-lives, whichever is longer, prior to randomisation.
20. Excessive use of alcohol (i.e. drink more than 2 standard units of alcohol per day or >8 standard units per week), including positive results for the alcohol breath test at Screening, Compliance Check, and Run-in/Randomization (Baseline) visits or is unwilling to abstain from alcohol consumption within 3 hours before bedtime for the duration of their participation in the study.
21. Recreational drug use, including positive results for the urine drugs of abuse test during at Screening, Compliance Check and Run-in/Randomization (Baseline) visits.
22. Use of any investigational drug or involvement in another clinical trial within 30 days of Screening.
23. Use of anti-coagulant drugs such as warfarin or those known to be metabolized by CYP450 enzymes, within 30 days of Screening.
24. Use of treatments for insomnia (e.g. cognitive-behavioral therapy and Central Nervous System-active drugs), within 30 days of Screening.
25. Self-reported or physician diagnosed comorbid nocturia resulting in frequent (>2) need to get out of bed to use the bathroom during the night.
26. Any history of a medical or psychiatric condition that, in the opinion of the Investigator, may affect the subject's safety or interfere with the study assessments.
27. Scheduled for major surgery during the study.
28. Shift work, jet lag or trans-meridian travel (three time zones) in the past month, at Screening and while on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Mean change from study baseline of insomnia severity index (ISI) score at 8 weeks | 8 weeks
  The insomnia severity index (ISI) is a seven-item self-report questionnaire used to assess the severity of the insomnia disorder.
  Total score ranges from 0-28. 0 - 7 No clinically significant insomnia. 8 - 14 Subthreshold insomnia. 15 - 21 Clinical insomnia (moderate severity) 22 - 28 Clinical insomnia (severe)
Mean change from study baseline in subject sleep efficiency (sSE) at 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Darren Mansfield, Principal Investigator — Monash Health
Locations (5):
- Australia (5):
  - Pioneer Clinical Research, North Sydney, New South Wales
  - Key Health, CBD South, Sydney, New South Wales
  - Griffith University, Southport, Queensland
  - Monash Health, Clayton, Victoria
  - Captain Stirling Medical Centre, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No